CLINICAL TRIAL: NCT03461718
Title: Ketamine as a Sedation Adjunct for Endoscopic Procedures
Brief Title: Ketamine for Endoscopic Sedation in Outpatient Adult Endoscopy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jerome Edelson, Physician, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2017.175
Record Dates: First submitted 2018-02-23; First posted 2018-03-12 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Administration and Dosage of Ketamine; Endoscopic Sedation
MeSH Terms: interventions — Ketamine; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Group will receive ketamine 0.5-1mg/kg for a loading dose then subsequent IV pushes of 10-20mg for maintenance. 1mg IV of midazolam will be administered prior to ketamine for anxiolysis and to help minimize emergence reaction.
  Interventions: Drug: Ketamine; Drug: Midazolam injection
- Control (Active Comparator): This group will receive midazolam and fentanyl alternated as currently preformed for endoscopy.
  Interventions: Drug: Midazolam injection; Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — Experimental arm for sedation.
  Arms: Ketamine
Drug: Midazolam injection — Part of standard sedation regimen and anxiolysis and for minimization of emergence reaction
Drug: Fentanyl — Part of standard sedation regimen
  Arms: Control

SUMMARY:
We will be investigating the use of ketamine in sedation for endoscopic procedures, specifically outpatient endoscopy including esophagoduodenoscopy (EGD) and colonoscopy. Participants will be randomized to one of two arms including conventional moderate sedation with midazolam and fentanyl or the ketamine arm. They will then undergo the planned procedure. Physicians preforming the procedure will be surveyed following the procedure and patients will be surveyed twice, once after meeting criteria for discharge on day of the procedure and a second time 48 hours following the procedure.

DETAILED DESCRIPTION:
In this study, the investigators plan to conduct a single blinded randomized controlled trial in the Gastroenterology Service to demonstrate the efficacy of ketamine and its utility in moderate sedation. Patients presenting to the endoscopy lab for esophagogastroduodenoscopy (EGD) and/or colonoscopy who meet inclusion criteria will be approached, and if amenable, will be consented and enrolled. Patients will be randomized to receive either a ketamine loading dose and then subsequent doses IV ketamine and midazolam 1mg IV prior to administration of ketamine or standard fentanyl/midazolam moderate sedation during their procedure. Participants will then undergo the planned procedure. The primary outcome will be patient satisfaction, which will be measured using the validated "Patient Satisfaction with Sedation" instrument (PSSI). A number of secondary outcomes will include the following: (1) provider satisfaction (measured using and the "Clinician Satisfaction with Sedation" instrument (CSSI), (2) the time from sedation administration to procedure start (when the scope is inserted), (3) the time from sedation to recovery (defined as the time from the end of the procedure until the patient meets discharge criteria from the recovery area), (4) time to cecum (for colonoscopy) total doses of medications given (midazolam, fentanyl, and ketamine), (5) overall time of the procedure, (6) adverse events, (7) changes in vital signs, (8) and the need for additional medications, in particular reversal agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 to 65 years who present to the GI clinic for an EGD or colonoscopy

Exclusion Criteria:

* Poor vital sign stability
* Hypoxia: O2 < 92%,
* Hypotension, hypertension, heart rate and respiratory rates greater than 20% above or below normal as dictated by normal ranges in SAMMC protocol
* Any allergy to ketamine, fentanyl, or midazolam
* Patient is pregnant or refuses pregnancy test, in women of child-bearing potential.*
* American Society of Anesthesiologists (ASA) score>3
* Presence of a history of psychosis, hallucinations, and/or a psychotic disorder
* History of increased intracranial pressure/ hypertensive hydrocephalus within the last 3 months
* Active pulmonary infection or disease.
* History of airway instability, tracheal surgery, or tracheal stenosis.

  * * Not applicable if patient is a female over 50 years old or has had a hysterectomy and/or oophorectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Provider satisfaction | Measured within 15 minutes post proceudre
  Measured with CSSI score. This consists of a questionnaire administered to the provider following the procedure with questions detailing different aspects of the procedure. Answers will be summed and the scores are normalized to a scale of 0-100 (high scores denote higher satisfaction).

SECONDARY OUTCOMES:
Sedation time | During the procedure
  Time from sedation administration until procedure start, will be measured in minutes
Time to cecum (for colonoscopy) | During the procedure
  Time required for endoscopist to reach the cecum, will be measured in minutes
Total dose of medications given | During the procedure
  All doses of medications will be summed and reported.
Overall procedure time | During the procedure
  The time from procedure start to procedure completion will be measured in minutes
Adverse events | During the procedure
  Are detailed in the protocol. We will be recording the presence or absence of adverse events.
Changes in vital signs | During the procedure
  As defined in the protocol. We will be recording all vital signs for later analysis.
Need for additional medications, ie reversal agents | During the procedure
  Will be measured as yes or no, specific dose and medication will be recorded for analysis.
Patient Satisfaction | After patient reaches criteria for discharge as listed above, a survey will be preformed. It will also be preformed 48 hours post procedure with the patients being called. Two surveys will end patient participation in the study.
  Measured with PSSI score. This consists of a questionnaire administered to the provider following the procedure with questions detailing different aspects of the procedure. Answers will be summed and the scores are normalized to a scale of 0-100 (high scores denote higher satisfaction). Criteria for discharge are at least 30 minutes elapsed since the last dose of sedative medication was administered, presence of protective reflexes (swallow and gag), stable vital signs, patient passes trial of ambulation (if was ambulating prior to procedure, a responsible adult is present to drive patient home and remain with the patient the length of two half-lives of the medications administered for sedation, and there are no staff concerns about safety. After the patient meets discharge criteria, a survey will be preformed. It will also be repeated once at the 48 hour post-procedure time. Conclusion of the two surveys concludes patient participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome C Edelson, MD, Principal Investigator — BAMC; John G Gancayco, MD, Study Chair — BAMC; Cyrus V Edelson, MD, Study Director — BAMC
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelson JC, Edelson CV, Rockey DC, Morales AL, Chung KK, Robles MJ, Marowske JH, Patel AA, Edelson SFD, Subramanian SR, Gancayco JG. Randomized Controlled Trial of Ketamine and Moderate Sedation for Outpatient Endoscopy in Adults. Mil Med. 2024 Jan 23;189(1-2):313-320. doi: 10.1093/milmed/usac183. PMID 35796486